CLINICAL TRIAL: NCT04869072
Title: A Phase i, Open-label, Single-centre Clinical Study to Evaluate Safety and Efficacy of Passive Immunization of High-risk SARS-CoV-2 Positive Patients With Convalescent Plasma Therapy
Brief Title: Convalescent Plasma Therapy - Zurich Protocol
Acronym: CPT-ZHP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00787
Record Dates: First submitted 2021-04-08; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-center, phase I study to assess the safety and efficacy of convalescent plasma therapy (CPT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Convalescent plasma — Convalescent plasma will be delivered as FFP. Three units of 200ml CP/FFP harvested from one donor will be transfused to one recipient, i.e. there will be a match between donor and recipient and each recipient will receive CP/FFP only from one donor.
  CP/FFP will be administered intravenously at the infusion rate of 100ml/hour, starting from day 0, with a new transfusion every 24 hours, for a total of 3 transfusions (see scheme).
  Other Names: Fresh Frozen Plasma (FFP)

SUMMARY:
This is an open-label, single-center, phase I study to assess the safety and efficacy of convalescent plasma therapy (CPT) obtained from donors who were tested positive for SARS-CoV-2 and fully recovered from the infection and administered to patients who are infected with the new coronavirus and present dyspnea or a poor prognosis

DETAILED DESCRIPTION:
The outbreak of a new highly contagious and life-threatening infective disease was first reported in China in December 2019. Regardless of the undertaken containing measures, its spreading could not be effectively stopped and currently we are confronting the pandemic diffusion of a newly identified Coronavirus (SARS-CoV-2) (1). This causes a systemic disease, known as (Coronavirus Disease-19) COVID-19, characterised by a broad spectrum of clinical manifestations, including ineffective hyper-inflammation and severe pneumonia, with provisional epidemiologic data indicating a mortality rate of 0.1-15% (2). Do to the lack of vaccination, specific anti-virus sera or monoclonal antibodies, the therapeutic efforts to limit COVID-19 mostly rely on the empirical use of anti-viral drugs. Therefore, being the option of an active immunisation not available and because of the controversial efficacy of the available anti-viral therapies (3), we suggest the option of a passive immunisation for those patients who are infected with the new coronavirus and present dyspnea or a poor prognosis. The use of convalescent plasma, i.e. plasma obtained from donors who were tested positive for SARS-CoV-2 and fully recovered from the infection, could provide a rapid protection, limiting the observed evolution of COVID-19 towards life-threating manifestations (7-9).

When carried on according to standardised measures, the transfusion of plasma is highly safe (10-11) and we assume that products containing anti- SARS-CoV- 2 antibodies will provide the recipients a passive immunity through different mechanisms, including viral neutralisation, antibody-dependent cellular cytotoxicity and/or phagocytosis.

ELIGIBILITY:
Inclusion Criteria:

A) Proven Sars-CoV-2 by PCR and hospitalization for COVID-19 in combination with either (1) or (2):

1. Age ≥50

   AND (at least one):
   * Pre-existing cardiovascular disease
   * Diabetic disease
   * Immunodeficiency/immunosuppression
   * Neoplastic disease
   * COPD or chronic liver disease or chronic renal failure
2. Age ≥18

AND (at least one):

* SpO2 ≤ 94% on room air or requiring supplemental oxygen at screening
* Typical changes on chest x-ray and/or lung-CT scan
* Immunosuppression or neoplastic disease

B) Informed Consent as documented by signature (Appendix Informed Consent Form) of the patient or, in case of inability, of the next relative/care-taking person. In the latter case, an independent doctor will also be involved and her/his signature will be required in order to enrol the patient.

Exclusion Criteria:

1. Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product (FFP)
2. Known IgA deficiency
3. Cytokine Release Syndrome grade ≥3 (see score)*
4. ARDS
5. Patients already hospitalized in intensive care unit and/or already receiving mechanical ventilation
6. Known or suspected non-compliance, drug or alcohol abuse
7. Previous enrolment into the current study
8. Enrolment of the investigator, his/her family members, employees and other dependent persons
9. Women who are pregnant or breast feeding
10. Intention to become pregnant during the course of the study
11. Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Please note that female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Safety of CPT applied to COVID-19 patients | clinical observation up to 48 hours after the last dose of plasma
  Absence of clinical signs of Transfusion Related Lung Inflammation (TRALI) and/or allergic reactions and/or Transfusion Associated Circulatory Overload (TACO)
Safety of CPT applied to COVID-19 patients | 1 week (laboratory monitoring up to 7 days after the last administration of plasma)
  Absence of laboratory signs of haemolytic reactions
Improvement of respiratory frequency | 3 weeks after the last administration of plasma
  Respiratory frequency will be measured at each study visit
Improvement of O2-saturation | 3 weeks after the last administration of plasma
  O2-Saturation will be measured at each study visit
Improvement of Inflammatory markers (C Reactive Protein, CRP) | 3 weeks after the last administration of plasma
  CRP will be measured at each study visit
Improvement of Inflammatory markers (Ferritin) | 3 weeks after the last administration of plasma
  Ferritin will be measured at each study visit
Improvement of Inflammatory markers (IL-6) | 3 weeks after the last administration of plasma
  IL-6 will be measured at each study visit
Improvement of coagulation-markers (D-dimer) | 3 weeks after the last administration of plasma
  D-Dimer will be measured at each study visit
Improvement of coagulation-markers (Fibrinogen) | 3 weeks after the last administration of plasma
  Fibrinogen will be measured at each study visit
Improvement of coagulation-markers (LDH) | 3 weeks after the last administration of plasma
  LDH will be measured at each study visit
Prevention of ICU-admission | 3 weeks after the last administration of plasma
  clinical conditions will be assessed throughout the study

SECONDARY OUTCOMES:
Characterisation of virus reaction to plasma Therapy | 10 Weeks
  Measurement of viral load after plasma therapy
Characterisation of the dynamic of humoral response after therapy | 10 Weeks
  Measurement of antibody-titres after plasma therapy
Better characterize the the in-vivo anti-virus humoral response against SARS-CoV-2. | 10 Weeks
  Performance of neutralisation assay after administration of plasma

CONTACTS AND LOCATIONS:
Overall Officials: Markus Manz, Professor, Study Chair — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marconato M, Abela IA, Hauser A, Schwarzmuller M, Katzensteiner R, Braun DL, Epp S, Audige A, Weber J, Rusert P, Schindler E, Pasin C, West E, Boni J, Kufner V, Huber M, Zaheri M, Schmutz S, Frey BM, Kouyos RD, Gunthard HF, Manz MG, Trkola A. Antibodies from convalescent plasma promote SARS-CoV-2 clearance in individuals with and without endogenous antibody response. J Clin Invest. 2022 Jun 15;132(12):e158190. doi: 10.1172/JCI158190. PMID 35482408